CLINICAL TRIAL: NCT06444035
Title: 35kDa Hyaluronan Fragment Injection Treatment Myofascial Pain Syndrome
Brief Title: Extended Therapeutic Effect of 35kDa Hyaluronan Fragment Injection in Patients With Chronic Pain Caused by Myofascial Pain Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nakhia Impex LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSHN005
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Chronic Wound; Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of myofascial pain syndrome by local injection of pain points (Experimental): Subjects received subcutaneous injection of HA35 injection 100mg / 5mL / day near the back pain point for 15 days.
  Interventions: Drug: HA35 injection

INTERVENTIONS:
Drug: HA35 injection — HA35/B-HA injection (Registration number L20200708MP07707; Ministry of Health). The subjects can continue to take oral analgesics during the treatment period, and the comparison of the dose and interval days of the analgesics before and after the treatment can also be used as the effect judgment of the injection.
  Other Names: B-HA injection

SUMMARY:
To verify the efficacy and safety of HA35 in chronic pain management and to further supplement effective treatments for chronic pain, we designed a proof-of-concept clinical study. This study aims to evaluate the 15-day treatment of HA35 on patients with myofascial pain syndrome and to observe the effects for up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, aged 18-65 years old ;
* suffering from muscle strain, sprain, fall, wind and other diagnosed as myofascitis in patients with chronic back pain;
* the pain reported by the subject should reach level 3 or higher on the digital rating scale of 0-10 ( 0 means no pain, 10 represents the strongest pain imaginable );
* the mental state is good, and the pain level can be evaluated independently;
* be able to cooperate with the treatment independently and sign a written consent.

Exclusion Criteria:

* Previous severe trauma with permanent musculoskeletal dysfunction;
* symptomatic lumbar disc herniation with neurological deficits;
* specific spinal diseases, including rheumatoid arthritis, ankylosing spondylitis, and osteoporosis;
* diagnosed with mental illness;
* agree not to sign the written consent;
* pregnant, lactating or fertile women;
* currently participating ( or participating in the past 30 days ) in research-based treatment or equipment trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Chronic myofascial pain score | after treatment 1 day, 3 days, 5 days, 15 days, 30 days, 60 days, 90 days
  Subjective measurements of pain were submitted using the Numerical Pain Rating Scale (NPRS). Scored at 0-10, the higher the score, the more obvious the pain.

SECONDARY OUTCOMES:
Overall pain assessment during injection therapy and follow-up | after treatment 15 days, 30 days, 60 days, 90 days
  The global pain scale (GPS) was used to assess the global pain. The total consists of 20 items, each rated on a scale from 0 to 10. The sum of the scores for all items is divided by 2 to obtain the total score. The higher the score, the more significant the pain and its impact.
Satisfaction survey of injection treatment | after treatment 90 days
  A questionnaire survey was conducted on patients using the Satisfaction with Medication Questionnaire ( TSQM 1.4 ). There are 4 subscales and 14 questions: the Effectiveness Scale (questions 1-3), the Side Effects Scale (questions 4-8), the Convenience Scale (questions 9-11), and the Overall Satisfaction Scale (questions 12-14). Each subscale is scored from 0 to 100, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Nahia Impex Llc, Ulaanbaatar, Mongolia